CLINICAL TRIAL: NCT00000746
Title: A Phase I, Multicenter, Randomized Trial to Evaluate the Safety and Immunogenicity of a Recombinant Vaccinia-HIV Envelope Vaccine (HIVAC-1e) in Combination With a Panel of Subunit Recombinant HIV Envelope Vaccines
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Purpose: Prevention
Other Study IDs: AVEG 008; AVEG Protocol 008; 10553 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-11-04 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
Keywords: Vaccines, Synthetic; Vaccinia Virus; Viral Vaccines; HIV-1; HIV Envelope Protein gp160; HIV Envelope Protein gp120; AIDS Vaccines; HIV Seronegativity; HIV Preventive Vaccine
MeSH Terms: conditions — HIV Infections; Vaccinia | interventions — HIVAC-1e; VaxSyn HIV-1 (gp160) vaccine

INTERVENTIONS:
Biological: rgp120/HIV-1 SF-2
Biological: Env 2-3
Biological: HIVAC-1e
Biological: gp160 Vaccine (MicroGeneSys)

SUMMARY:
Primary: To determine in healthy volunteers whether priming with a vaccinia HIV-1 gp160 envelope gene recombinant vaccine (HIVAC-1e) followed by boosting with one of two subunit recombinant HIV-1 envelope vaccines (Env 2-3 and gp120) provides enhanced immunogenicity compared to vaccination with the gp120 subunit vaccine alone. (Per 10/01/92 amendment, boosts with VaxSyn (gp160) were eliminated.) To evaluate the immunogenicity of one versus two priming doses of HIVAC-1e prior to a boost with gp120. To compare the relative immunogenicity of the three subunit vaccines when administered as boosters.

Secondary: To examine the safety of administering the individual subunit vaccines in combination with HIVAC-1e and the safety of administering the gp120 subunit vaccine alone.

In a previous study of candidate HIV vaccines, the evidence suggested that administration of a booster vaccination with a different vaccine preparation may produce a better immune response than administration of HIVAC-1e vaccine alone.

DETAILED DESCRIPTION:
In a previous study of candidate HIV vaccines, the evidence suggested that administration of a booster vaccination with a different vaccine preparation may produce a better immune response than administration of HIVAC-1e vaccine alone.

Seventy healthy volunteers are randomized to one of four groups. Groups A and D receive one initial immunization with HIVAC-1e followed by two boosts with subunit gp120 and Env 2-3, respectively, at months 8 and 12. Group B receives two immunizations with HIVAC-1e at months 0 and 8 followed by a single boost with subunit gp120 at month 12. Group C receives three doses of subunit gp120 only at months 0, 8 and 12. (Per 10/01/92 amendment, boosts with VaxSyn (gp160) have been eliminated.) Subjects are followed for 18 months.

ELIGIBILITY:
Inclusion Criteria

Subjects must have:

* Normal history and physical exam.
* Negative HIV screening by ELISA, Western blot, and p24 antigen (PBMC HIV culture or HIV-specific PCR can be substituted for Western blot and p24 antigen).
* History of smallpox vaccination more than 5 years prior to enrollment.
* Normal urinalysis.
* Absolute CD4 count = or > 500 cells/mm3.

Prior Medication: Required:

* Vaccinia (smallpox) vaccination more than 5 years prior to study enrollment. Identifiable high-risk behavior for HIV infection as determined by screening questionnaire/interview.

Exclusion Criteria

Co-existing Condition:

Subjects with the following symptoms or conditions are excluded:

* Household contacts who are pregnant, < 12 months of age, have eczema, or have immunodeficiency disease or who use immunosuppressive medications.
* Hepatitis B surface antigenemia.
* Medical or psychiatric condition or occupational responsibilities that preclude compliance.

Subjects with the following prior conditions are excluded:

* History of immunodeficiency or chronic illness.
* Eczema within the past year.

Prior Medication:

Excluded:

* Prior experimental HIV vaccine.
* Immunoglobulin administration or use of experimental agent within the past 2 months.
* History of immunosuppressive medications.

Prior Treatment:

Excluded:

* Blood or blood product transfusion within the previous 6 months.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56
Dates: Study Completion 1994-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey L, Study Chair
Locations (1):
- JHU AVEG, Pittsburgh, Pennsylvania, United States

REFERENCES:
- [Background] Clements ML, Corey L, Weinhold K, Schwartz D, Siliciano R, Matthews T, Hsieh R, Graham B, Keefer M, Gorse G, Zolla-Pazner S, Mascola J, Duliege A, Excler J, Tartaglia J, Paoletti E, Hu SL. HIV immunity induced by priming with canarypox or vaccinia-gp160 recombinants and boosting with rgp120. Inst of Hum Virol Annu Meet. 1996 Sept 7-13
- [Background] Graham BS, Belshe RB, Clements ML, Dolin R, Corey L, Wright PF, Gorse GJ, Midthun K, Keefer MC, Roberts NJ Jr, et al. Vaccination of vaccinia-naive adults with human immunodeficiency virus type 1 gp160 recombinant vaccinia virus in a blinded, controlled, randomized clinical trial. The AIDS Vaccine Clinical Trials Network. J Infect Dis. 1992 Aug;166(2):244-52. doi: 10.1093/infdis/166.2.244. PMID 1353102